CLINICAL TRIAL: NCT04531527
Title: HT201308- Human Phototoxicity Test
Brief Title: Study to Learn More About the Potential of Antifungal Cream V61-044 Containing Trolamine to Cause Irritant Reaction of the Skin to Ultra Violet Light in Healthy Human Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18154
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Dermatitis, Phototoxic
MeSH Terms: conditions — Dermatitis, Phototoxic | interventions — butenafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phototoxicity reaction test (Experimental): Participants received approximately 60 μl of Butenafine HCl 1% on the treated irradiated test site followed by Ultraviolet Radiation (UV) irradiation and to the treated non-irradiated test site without UV irradiation. Participants also had two more test sites, the untreated irradiated control site without Butenafine HCl 1% followed by UV irradiation and the untreated non-irradiated control site without Butenafine HCl 1% or UV irradiation. All test sites were evaluated for erythema on the following day. Afterwards, participants received same procedure on all 4 test sites, and evaluation of the test sites occurred at 24 hours and 48 hours post-irradiation.
  Interventions: Drug: Butenafine HCl 1% (BAY1896425)

INTERVENTIONS:
Drug: Butenafine HCl 1% (BAY1896425) — Approximately 60 μl of Butenafine HCl 1% applied twice to the treated irradiated site and to the treated non-irradiated site for a total application of 240 μl of Butenafine HCl 1%.
  Other Names: Antifungal Cream V61-044 containing Trolamine

SUMMARY:
In this study researchers want to gather information about the potential of Antifungal Cream V61-044 containing Trolamine to produce a phototoxic reaction on the skin. A phototoxic reaction is an irritant reaction of the skin to ultra violet light. In order to find this out the study drug will be applied to the skin of healthy human subjects. By using a solar simulator to generate a UV spectrum similar to that of sunlight the potential of the study drug to produce a superficial reddening of the skin will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been between the ages of 18 and 60 years;
* Participants must have been lightly pigmented (Fitzpatrick skin phototypes I, II, III);
* Participants must have been in good general health as determined by the subject's medical history;
* Participants must have been willing to avoid tanning bed usage and additional sun exposure during the trial and follow-up period;
* Participants must have been willing to refrain from using any new topical products during the trial;
* Participants must have been able and willing to cooperate with the Investigator and research staff, to have test materials applied according to protocol, and to complete the full course of the trial;
* Participants must have been willing to report any medications taken during the trial and refrain from taking any medications during the trial that might produce photoreactions;
* If female, participants must produce a negative urine pregnancy test prior to the initiation and also at the completion of the trial.

Exclusion Criteria:

* Participants must not have had visible sunburn;
* Participants must not have had a history of sun hypersensitivity/photosensitivity, or photosensitive dermatoses;
* Participants must not have had a history of allergies or sensitivities to cosmetics, toiletries, or any dermatological products;
* Participants must not have recently used any systemic or topical drugs which could have caused a photoreaction or may have interfered with the trial;
* Participants must not have had any known skin conditions that might interfere with the proper conduct of the trial;
* Participants must not have had scars, moles, excessive hair, or other blemishes over the mid or lower back which might have interfered with the test or the grading of the test sites;
* Participants must not have had significant history of internal disease that may have interfered with the evaluation of the test material as determined by the Investigator;
* Participants must not have been pregnant, planning pregnancy, or nursing a child during the trial period;
* Participants must not have used a tanning bed or other artificial tanning lights within the past two months;
* Participants must not have participated in a patch test involving the back within four weeks prior to the start of the trial;
* Participants must not have concurrently participated in any other clinical or consumer test;
* Participants must not have had other conditions considered by the Investigator as sound reasons for disqualification from enrollment into the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2013-06-28 (Actual); Study Completion 2013-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Fairfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at single center in the US, between 24 JUN 2013 (first subject first visit) and 28 JUN 2013 (last subject last visit).
Pre-assignment Details: A total of 32 subjects were enrolled in the study and 29 received study treatment.
Groups:
- Phototoxicity Reaction Test: Participants received approximately 60 μl of Butenafine HCl 1% on the treated irradiated test site followed by UV irradiation and to the treated non-irradiated test site without UV irradiation. Participants also had two more test sites, the untreated irradiated control site without Butenafine HCl 1% followed by UV irradiation and the untreated non-irradiated control site without Butenafine HCl 1% or UV irradiation. All test sites were evaluated for erythema on the following day. Afterwards, participants received same procedure on all 4 test sites, and evaluation of the test sites occurred at 24 hours and 48 hours post-irradiation.
Period: Overall Study
Arm/Group | Phototoxicity Reaction Test
Started | 32
Treated | 29
Completed | 29
Not Completed | 3
Not completed — Found to be Ineligible | 3

BASELINE CHARACTERISTICS:
Arm/Group | Phototoxicity Reaction Test
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 27
  Hispanic | 3
  Caucasian/African American | 1
  Caucasian/Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Phototoxic Reaction Evaluation Reported as Number of Test Site With Different Erythema Score
Description: Evaluation of the test sites after irradiation used following scoring system: score 0=Normal skin; score 1=Faint, barely perceptible to moderate redness with poorly defined margins (not clinically significant); score 2=Moderate to intense redness with well defined margins; score 3=Redness plus well defined edema; score 4=Redness plus papules, vesicles, or ulceration. All four test sites were evaluated for gross changes according to the Erythemal Scoring Scale and if necessary the Additional Scoring system immediately before irradiation, 24 hours after irradiation, and 48 hours after irradiation (3 different time points), thus for each type of test site (i.e. treated irradiated test site), a total of 87 test sites with scores were collected (i.e., 29 participants *3 time points = 87 sites).
Time Frame: Immediately before irradiation, 24 hours after irradiation, and 48 hours after irradiation
Population: Subjects who received treatment
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Phototoxicity Reaction Test
Number analyzed (Participants) | 29
Number analyzed (Test site) | 87
Test site
  Treated irradiated test site, score=0 | 77
  Treated irradiated test site, score=1 | 10
  Treated non-irradiated test site, score=0 | 85
  Treated non-irradiated test site, score=1 | 2
  Untreated irradiated test site, score=0 | 78
  Untreated irradiated test site, score=1 | 9
  Untreated non-irradiated test site, score=0 | 85
  Untreated non-irradiated test site, score=1 | 2

2. Secondary Outcome: Development of Erythema on the Treated Non-irradiated Test Sites, Which Would Indicate Irritant Contact Dermatitis and a Pre-existing Allergic Contact Dermatitis
Description: as for outcome 1
Time Frame: Immediately before irradiation, 24 hours after irradiation, and 48 hours after irradiation
Population: Subjects who received treatment
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Phototoxicity Reaction Test
Number analyzed (Participants) | 29
Number analyzed (Test site) | 87
Test site
  Treated non-irradiated test site, score=0 | 85
  Treated non-irradiated test site, score=1 | 2

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | Phototoxicity Reaction Test
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No information based on the conduct of the study (incl. protocol, data resulting from the study, or the fact that the study was being conducted) will be released without prior written consent of the sponsor unless the requirement is superseded by State or Federal law.